CLINICAL TRIAL: NCT06488547
Title: Musculoskeletal Disorders and Stress Management, in Employees
Brief Title: Stress and Musculoskeletal Health in Employees
Acronym: MUStress
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Collaborators: THE ENDOCRINE UNIT OF THE UNIVERSITY OF ATHENS (Unknown)
Responsible Party: Principal Investigator, Eleni Zigkiri, PhD (c), University of Thessaly
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2224/14-04-2022
Record Dates: First submitted 2024-06-13; First posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-06

CONDITIONS: Musculoskeletal Diseases or Conditions; Musculoskeletal Pain; Musculoskeletal Health; Stress; Work Related Stress; Occupation-related Stress Disorder; Medically Unexplained Symptoms
Keywords: stress management; stress biomarkers; musculoskeletal health; work-related; biofeedback; saliva cortisol; HRV
MeSH Terms: conditions — Musculoskeletal Diseases; Musculoskeletal Pain; Occupational Stress; Medically Unexplained Symptoms | interventions — Autogenic Training

STUDY DESIGN:
Intervention Model Description: interventional group and control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stress Managemenet Group (Experimental): Participants will be instructed and trained with two stress management techniques (Diaphragmatic Breathing- DB and Progressive Muscle Relaxation-PMR), along with biofeedback training in diaphragmatic breathing.
  During the eight weeks of the program, participants in the intervention group will receive information regarding stress, work-related stress factors, musculoskeletal health and disorders, the Medically Unexplained Symptoms-MUS, occupational psychosocial hazards, lifestyle habits (healthy diet, sedentary life, sleep, hygiene).
  Moreover, participants will be informed about how to manage stress related factors at the workplace, and its symptoms, through lifestyle modifications along with ergonomic guidance at work and in relation with their musculoskeletal health, the psychosocial hazards at work and their body response to work-related stress.
  Interventions: Other: Diaphragmatic breathing (DF); Other: Progressive Muscle Relaxation (PMR)
- Control Group-CG (No Intervention): Participants will receive only information regarding ergonomic practices and tips able to be appilied at the workplace.

INTERVENTIONS:
Other: Diaphragmatic breathing (DF) — Diaphragmatic breathing (DF), also known as belly or abdominal breathing, is a technique that can teach people how to use their diaphragm correctly while breathing, in order to activate the parasympathetic branch of the autonomic nervous system and to control stress.
  Arms: Stress Managemenet Group
Other: Progressive Muscle Relaxation (PMR) — Progressive Muscle Relaxation (PMR) is a technique that is helpful in the reduction of stress.
  PMR by alternately tensing and relaxing different muscle groups in the body helps participants to become more aware of physical sensations and can be particularly helpful to muscle tension and relaxation.
  Arms: Stress Managemenet Group

SUMMARY:
This study aims to evaluate potential correlation of stress as estimated by certain biological markers, namely saliva cortisol, Heart rate variability (HRV), Electromyography (EMG) with musculoskeletal system health status, and assess the impact of a stress management intervention..The intervention group will be trained to apply two evidence based stress management techniques and they will be guided with tips and advice about musculoskeletal health.

Impact of the intervention upon measured stress related markers will be assessed.

DETAILED DESCRIPTION:
The goal of this non-pharmacological randomized interventional study is to investigate work-related stress in relation to the musculoskeletal health of employees.

The primary purpose of this study is to investigate if stress management interventions in employees can improve self-reported musculoskeletal health problems or Medically Unexplained Symptoms (MUS), in relation with biomarkers of stress.

Secondary outcomes will include quality of life improvement and the number of absences from work, due to musculoskeletal conditions.

The main question aims to answer if specific stress management techniques can improve the self-reported musculoskeletal health of employees.

Researchers will compare the results between two groups (one participating in the the six (6) week program and the other not participating) to measure the effect size in the intervention group and between groups.

Participants from both groups will be measured twice (on week 1 and week 8) with the same self-report questionnaires and stress biomarkers, if possible. Especially for the intervention group a six-week stress management program will be applied. This will include the participation in one and a half hour consultation meetings about stress, musculoskeletal health, psychosocial work-related factors, and how to improve well-being and work/life satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Writing and reading greek.
* Consent to provide their medical history.
* Consent to be measured with electronic devices.

Exclusion Criteria:

* Employees who are close to retirement (at least 2 years before) and those for whom any known factor may prevent them from completing the intervention (eg travel, transfer).
* Pregnancy.
* Pacemaker, history of seizures.
* Diagnosed musculoskeletal injury.
* Diagnosed diseases such as: osteoarthritis, autoimmune diseases (rheumatoid arthritis, lupus, etc.), stroke, myocardial infarction, malignant neoplasms, psychiatric disease, disability.
* Systematic reception of cortisone and anti-inflammatory treatment, up to at least three months before the intervention.
* Drugs or substances.
* Participation in another interventional program of musculoskeletal rehabilitation, physical therapy, stress management or health promotion.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Heart Rate Variability (HRV) | 8 weeks
  Heart Rate Variability (HRV) has been widely used as an indicator for work-related stress. It measures the variation in time between each heartbeat and is controlled by the autonomic nervous system.
Saliva cortisol | 8 weeks
  Salivary cortisol has been used as an indicator for stress. Pre-post intervention differences between diurnal circadian rhythm in the saliva cortisol of the participants will be measured, in order to evaluate the efficiency of the intervention upon homeostatic load.
Musculoskeletal symptoms | 8 weeks
  Musculoskeletal symptoms will be assessed with the Nordic Musculoskeletal Questionnaire (NMQ). NMQ is a standardized questionnaire for the assessment of musculoskeletal problems in nine different body regions (neck, shoulders, upper back, elbows, wrist/hands, lower back, hips/thighs, knees, ankles/feet). General questions include 40 forced-choice items where responders could indicate if they had musculoskeletal problems (aches, pain, discomfort) in the last 12 months or seven days. Additional questions ask the participants to report if the musculoskeletal problems had led to inability to perform daily tasks and normal activities.
  Work-related stress can lead to physical strain, which in turn can lead to musculoskeletal tension and disorders. Musculoskeletal disorders (MSDs) are a common type of occupational diseases and have become the main cause of absenteeism and early retirement in the working population.

SECONDARY OUTCOMES:
Sort Form Health Survey questionnaire (SF-36) | 8 weeks
  Quality of life will be measured with the Short Form survey (SF-36) self-report questionnaire. SF-36 provides comprehensive information of an individual health status and assesses eight domains of health such as: Physical functioning, Role limitations due to physical health, Role limitations due to emotional problems, Energy/ fatigue (vitality), Emotional wellbeing, Social functioning, Pain, and General health. It provides valuable insights into participants' perceived health status and overall quality of life. All questions are scored on a scale from 0 to 100, reflecting a range from lowest to highest possible quality of life.
  Scoring the SF-36 involves a two-step process. At first each question must be pre- coded with a numeric value which is then recorded according to a scoring key and then the second step involves averaging the recorded values from items within the same scale to compute the total scale score.

OTHER OUTCOMES:
Phychosocial work-related stress | 8 weeks
  Psychosocial work-related stress factors will be measured with the Copenhagen Psychosocial Questionnaire (COPSOQ-II medium version). The medium version of the questionnaire consists of 8 domains, 28 dimensions and 87 items. Each item scores from 0-100 (i.e. 0, 25, 50, 75, and 100 for a five response category item). The scale score is computed as the mean item score. Higher total score indicates that the employee experiences greater work-related psychosocial risk factors.
Perceived Stress | 8 weeks
  Perceived stress will be measured with the Perceived Stress Scale (PSS-14), which is a self-report questionnaire with 14 items. It measures the perception of stressful experiences of the responder by rating the frequency of the feelings and thoughts related to events over the past month. Between items half of them are considered negative and the other as positive. Each answer responds on a five point Likert-type scale (0-never to 4=very often). Total score ranges from 0-56 and higher scores indicate greater perceived stress.
Depression - Anxiety - Stress | 8 weeks
  Depression, Anxiety and Stress parameters will be measured with the Depression Anxiety Stress Scales (DASS-21), which is a self-reported questionnaire designed to measure the emotional states of depression, anxiety and stress. It consists of three subscales of depression, anxiety and stress. Each subscale consists of seven items which are answered on a 4-point Likert-type scale. the answers ranging from 0 ("does not apply to me at all") to 3 ("applies to me very much") scales. The score of each subscale has to be multiplied by 2 to obtain the total subscale scores. The total scores of each subscale range from 0 to 42 points, with higher scores indicating more severe depression/anxiety/stress symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Eleni Zigkiri, PhD (c), Principal Investigator — University of Thessaly
Locations (2):
- Greece (2):
  - University of Thessaly, Larissa, Biopolis- Larissa
  - The Endocrine Unit of the University of Athens, Athens

REFERENCES:
- [Result] Nakao M. Work-related stress and psychosomatic medicine. Biopsychosoc Med. 2010 May 26;4(1):4. doi: 10.1186/1751-0759-4-4. PMID 20504368
- [Result] Goessl VC, Curtiss JE, Hofmann SG. The effect of heart rate variability biofeedback training on stress and anxiety: a meta-analysis. Psychol Med. 2017 Nov;47(15):2578-2586. doi: 10.1017/S0033291717001003. Epub 2017 May 8. PMID 28478782
- [Result] Lehrer PM, Gevirtz R. Heart rate variability biofeedback: how and why does it work? Front Psychol. 2014 Jul 21;5:756. doi: 10.3389/fpsyg.2014.00756. eCollection 2014. PMID 25101026
- [Result] Eatough EM, Way JD, Chang CH. Understanding the link between psychosocial work stressors and work-related musculoskeletal complaints. Appl Ergon. 2012 May;43(3):554-63. doi: 10.1016/j.apergo.2011.08.009. Epub 2011 Sep 23. PMID 21944295
- [Result] Buscemi V, Chang WJ, Liston MB, McAuley JH, Schabrun SM. The Role of Perceived Stress and Life Stressors in the Development of Chronic Musculoskeletal Pain Disorders: A Systematic Review. J Pain. 2019 Oct;20(10):1127-1139. doi: 10.1016/j.jpain.2019.02.008. Epub 2019 Feb 22. PMID 30797962
- [Result] Maina G, Palmas A, Bovenzi M, Filon FL. Salivary cortisol and psychosocial hazards at work. Am J Ind Med. 2009 Mar;52(3):251-60. doi: 10.1002/ajim.20659. PMID 19023870
- [Result] Wang J, Zhu L, Song L, Zhou Z, Chan W, Li G, Zhou L, Xiao J, Lian Y. A cohort study on the association between changing occupational stress, hair cortisol concentration, and hypertension. PLoS One. 2023 May 17;18(5):e0285623. doi: 10.1371/journal.pone.0285623. eCollection 2023. PMID 37196014